CLINICAL TRIAL: NCT02239536
Title: Hot Snare Polypectomy Vs. Hot Snare Polypectomy After Saline Injection for the Complete Resection of Neoplastic Colorectal Polyps: Prospective, Randomized Controlled Trial
Brief Title: Hot Snare Versus Hot Snare Polypectomy With Saline Injection for Colorectal Polyps
Acronym: HSPvsHSPASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bo-In Lee (Other)
Collaborators: St Vincent's Hospital (Other); Incheon St.Mary's Hospital (Other)
Responsible Party: Sponsor-Investigator, Bo-In Lee, MD, PhD, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC14TIMI0039K
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Polyp of Large Intestine
Keywords: neoplastic colorectal polyp; hot snare polypectomy; hot snare polypectomy after saline injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hot snare polypectomy (Experimental): Intervention: Procedure: removal of eligible polyps using hot snare polypectomy technique
  Interventions: Procedure: hot snare polypectomy
- Hot snare polypectomy(saline injection) (Experimental): Intervention: Procedure: removal of eligible polyps using hot snare polypectomy after saline injection technique
  Interventions: Procedure: hot snare polypectomy after saline injection

INTERVENTIONS:
Procedure: hot snare polypectomy — hot snare polypectomy using electrosurgical snare with application of electrocautery for eligible polyps
  Arms: Hot snare polypectomy
Procedure: hot snare polypectomy after saline injection — hot snare polypectomy after saline injection using electrosurgical snare with application of electrocautery for eligible polyps
  Arms: Hot snare polypectomy(saline injection)

SUMMARY:
The complete removal of colorectal polyp is required to prevent tumor recurrence and development of potential interval cancers. However, several studies have shown high incomplete resection rate in endoscopic removal of neoplastic colorectal polyps larger than 5 mm. The polypectomy techniques using hot snare are usually used for the removal of these polyps. However, the optimal technique for complete resection of these polyps is unknown. There are few data comparing hot snare polypectomy with hot snare polypectomy after saline injection for complete resection of colorectal polyps (5mm or larger). The aim of this study is to compare hot snare polypectomy with hot snare polypectomy after saline injection for removal of 5-10mm sized colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 30
* 5~10mm sized colorectal polyps
* Informed consent

Exclusion Criteria:

* Inflammatory bowel diseases (Crohn's disease, or ulcerative colitis)
* Patient undergoing antiplatelets (aspirin, clopidogrel and others) or anticoagulant therapy
* ASA class III or more
* Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if he/she were to participate in the study

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo-In Lee, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Division of Gastroenterology; Seoul St. Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dwyer JP, Tan JYC, Urquhart P, Secomb R, Bunn C, Reynolds J, La Nauze R, Kemp W, Roberts S, Brown G. A prospective comparison of cold snare polypectomy using traditional or dedicated cold snares for the resection of small sessile colorectal polyps. Endosc Int Open. 2017 Nov;5(11):E1062-E1068. doi: 10.1055/s-0043-113564. Epub 2017 Oct 27. PMID 29250580
- [Background] Kim JS, Lee BI, Choi H, Jun SY, Park ES, Park JM, Lee IS, Kim BW, Kim SW, Choi MG. Cold snare polypectomy versus cold forceps polypectomy for diminutive and small colorectal polyps: a randomized controlled trial. Gastrointest Endosc. 2015 Mar;81(3):741-7. doi: 10.1016/j.gie.2014.11.048. PMID 25708763
- [Background] Kawamura T, Takeuchi Y, Asai S, Yokota I, Akamine E, Kato M, Akamatsu T, Tada K, Komeda Y, Iwatate M, Kawakami K, Nishikawa M, Watanabe D, Yamauchi A, Fukata N, Shimatani M, Ooi M, Fujita K, Sano Y, Kashida H, Hirose S, Iwagami H, Uedo N, Teramukai S, Tanaka K. A comparison of the resection rate for cold and hot snare polypectomy for 4-9 mm colorectal polyps: a multicentre randomised controlled trial (CRESCENT study). Gut. 2018 Nov;67(11):1950-1957. doi: 10.1136/gutjnl-2017-314215. Epub 2017 Sep 28. PMID 28970290
- [Derived] Kim SJ, Lee BI, Jung ES, Kim JS, Jun SY, Kim W, Ham H, Kim M, Lee SH, Lee HH, Park JM, Choi MG. Hot snare polypectomy versus endoscopic mucosal resection for small colorectal polyps: a randomized controlled trial. Surg Endosc. 2021 Sep;35(9):5096-5103. doi: 10.1007/s00464-020-07994-7. Epub 2020 Sep 28. PMID 32989532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were excluded if they have (1) a bleeding tendency or ever taken antiplatelet or anticoagulation therapy within 1 week before undergoing the procedure, (2) An inflammatory bowel disease, (3) a polyposis syndrome, or (4) an inability to provide informed consent.
Period: Overall Study
Arm/Group | Hot Snare Polypectomy | Hot Snare Polypectomy(Saline Injection)
Started | 190 | 172
Completed | 167 | 155
Not Completed | 23 | 17
Not completed — Non-neoplastic polyp | 23 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hot Snare Polypectomy | Hot Snare Polypectomy(Saline Injection) | Total
Number analyzed (Participants) | 167 | 155 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.7) | 63.0 (10.8) | 62.9 (10.7)
Sex/Gender, Customized [Number; unit: participants]
  Male | 114 | 98 | 212
  Female | 53 | 57 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 167 | 155 | 322
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 167 | 155 | 322
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Resection Rate
Description: Complete resection was defined as the absence of residual polyp in the resection margin
Time Frame: 2 weeks after
Measure: Count of Participants; unit: Participants
Arm/Group | Hot Snare Polypectomy | Hot Snare Polypectomy(Saline Injection)
Number analyzed (Participants) | 167 | 155
Participants
  Complete resection | 161 | 148
  Incomplete resection | 6 | 7
Statistical Analysis 1: Comparison: Hot Snare Polypectomy vs Hot Snare Polypectomy(Saline Injection); Test type: Other; p = 0.05, Chi-squared

2. Secondary Outcome: Lateral Margin
Description: Observation of maring on a recsected specimen
Time Frame: 2 weeks after
Measure: Count of Participants; unit: Participants
Arm/Group | Hot Snare Polypectomy | Hot Snare Polypectomy(Saline Injection)
Number analyzed (Participants) | 167 | 155
Participants
  Negative | 83 | 116
  Positive | 3 | 2
  Inconclusive | 91 | 37
Statistical Analysis 1: Comparison: Hot Snare Polypectomy vs Hot Snare Polypectomy(Saline Injection); Test type: Other; p = 0.05, Chi-squared
Statistical Analysis 2: Comparison: Hot Snare Polypectomy vs Hot Snare Polypectomy(Saline Injection); Test type: Other; p = 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 weeks after polypectomy
Description: Post-polypectomy bleeding was classified two categories, immediately bleeding defined as over 30 seconds continuous bleeding episode requiring any form of endoscopic hemostasis and delayed bleeding defined as between 24 hours and 2weeks after polypectomy requiring any form of endoscopic hemostasis (i.e. epinephrine injection, clipping or coagulation).
Arm/Group | Hot Snare Polypectomy | Hot Snare Polypectomy(Saline Injection)
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/155
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/155
Other Adverse Events (participants affected / at risk) | 17/167 | 13/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hot Snare Polypectomy (N=167) | Hot Snare Polypectomy(Saline Injection) (N=155)
Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) — Situations that require surgical treatment due to mucosal defects
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hot Snare Polypectomy (N=167) | Hot Snare Polypectomy(Saline Injection) (N=155)
Immediate bleeding (Gastrointestinal disorders) | 17 (17) | 12 (12) — continuous bleeding over 30 seconds requiring any form of endoscopic hemostasis (epinephrine injection, clipping or coagulation)
Delayed bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) — bleeding from the post-polypectomy site between 24 hours and 2 weeks after polypectomy
Post-polypectomy syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT02239536/Prot_SAP_000.pdf